CLINICAL TRIAL: NCT04993027
Title: Topical Vancomycin for Infection Prophylaxis in Total Hip and Knee Arthroplasty
Brief Title: Topical Vancomycin for Infection Prophylaxis in TJA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alberta Hip and Knee Clinic (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Principal Investigator, Nicholas Desy, Clinical Assistant Professor, Alberta Hip and Knee Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REB21-0490
Record Dates: First submitted 2021-05-13; First posted 2021-08-06 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Infection of Total Hip Joint Prosthesis; Infection of Total Knee Joint Prosthesis
MeSH Terms: interventions — Vancomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vancomycin Group: (Experimental): patients will have single dose of 1g vancomycin powder placed on their incision during surgery in addition to: pre- and post-operative intravenous antibiotic administration, sterile surgical helmet systems, saline pulse lavage irrigation, and antimicrobial drapes.
  Interventions: Drug: Vancomycin Powder
- Control Group (No Intervention): pre- and post-operative intravenous antibiotic administration, sterile surgical helmet systems, saline pulse lavage irrigation, and antimicrobial drapes.

INTERVENTIONS:
Drug: Vancomycin Powder — Vancomycin is a bactericidal aminoglycoside antibiotic which inhibits cell wall synthesis. It is effective against gram positive bacteria. Though most commonly administered intravenously, it can be delivered orally or directly into surgical incisions and wounds in certain indications.
  Other Names: Vancomycin Hydrochloride
  Arms: Vancomycin Group:

SUMMARY:
11% of the general population undergo total hip arthroplasty (THA) in their lifetime and 7% undergo total knee arthroplasty (TKA), with these rates expected to rise up to 50% by 2026. Periprosthetic joint infection (PJI) remains one of the most common complications, accounting for 30% of THA/TKA revision surgeries. Topical delivery of antibiotic powder may reduce the incidence of PJI but its potential drawbacks include wound healing complications, reduced osteoblast activity, third body wear, and antibiotic resistance. In THA and TKA, topical administration of vancomycin powder for the primary prevention of PJI has been studied in observational studies, but conclusions are limited due to the low incidence of PJI and high number of patients required to detect a significant difference. Investigators therefore propose a randomized controlled trial (RCT) investigating the impact of topical vancomycin compared to standard care on PJI rates following THA and TKA.

Aim: To determine whether topical vancomycin is a safe and effective intervention for the primary prevention of PJI after THA and TKA.

Study Design: This is a pilot multi-centre RCT to evaluate the study design and assess feasibility prior to implementation across Canada. Investigators aim to recruit 50 THA and 50 TKA patients.

Inclusion Criteria THA or TKA Patients aged 18 years or older Patients must complete 1 year follow-up Exclusion Criteria Patients undergoing surgery for inflammatory arthritis, post-traumatic arthritis, or avascular necrosis History or septic arthritis based on history or synovial aspirate Prior major operation on the affected joint Current immunosuppressive medications Vancomycin allergy or history of a vancomycin-related complication Recruitment: surgeons introduce study to the patients, research staff will conduct recruitment.

Intervention: Patients will be randomized preoperatively and remain blinded to their treatment arm. Patients allocated to the control group will have all standard care infection prophylaxis interventions. Patients allocated to the vancomycin group will undergo all the standard care measures in addition to 1g of powdered vancomycin applied to the wound.

Follow-up: Patients will complete follow-up at 2 weeks, 6 weeks, 3 months, 6 months, and 1 year visits.

Primary outcome: PJI in the same joint. Secondary outcome: PJI in THA and TKA subgroups:

Reoperation on the same joint Superficial and non-infectious wound complications All complications

DETAILED DESCRIPTION:
Hip and knee arthroplasty are the third and second most performed inpatient surgeries, respectively. Eleven percent of the general population undergo total hip arthroplasty (THA) in their lifetime and 7% undergo total knee arthroplasty (TKA), with these rates expected to rise up to 50% by 2026. Unfortunately, periprosthetic joint infection (PJI) remains one of the most common and devastating complications of hip and knee arthroplasty, accounting for 30% of revision surgeries.The incidence of PJI ranges from 0.2-1.6% for primary THA and 1-2% for primary TKA. Patients with PJI are subjected to repeated hospitalization and revision surgeries, which leads to increased morbidity and mortality as well as decreased functional outcomes. An estimated $1.6 billion USD is spent on treating hip and knee PJI in the United States yearly.

Topical delivery of antibiotic powder is a simple intervention which may reduce the incidence of PJI. Direct delivery of antibiotics to a target area allows for high local drug concentrations while limiting systemic side effects.Potential drawbacks of topical antibiotics include wound healing complications, reduced osteoblast activity, third body wear, and contribution to antibiotic resistance. Though systemic absorption is reduced, complications such as anaphylaxis, nephrotoxicity, and ototoxicity remain possible. Topical, intrawound administration of vancomycin powder has been well studied in spinal surgery for the prevention of surgical site infections (SSI), with good results. Based on this literature, vancomycin powder has been investigated for the prevention of SSI in multiple orthopaedic domains. In THA and TKA, topical administration of vancomycin powder for the primary prevention of PJI has been studied in a number of recent observational studies, but conclusions are limited due to the low incidence of PJI and high number of patients required to detect a significant difference.

Investigators have completed a systematic review meta-analysis of nine comparative observational studies investigating topical vancomycin for the primary prevention of PJI after hip and knee arthroplasty. Patients treated with topical vancomycin had a lower incidence of PJI compared to the control group (0.6% versus 1.8%, OR 0.40, p = 0.003). Excluding revision cases, patients undergoing primary hip or knee arthroplasty also had a lower incidence of PJI after topical vancomycin (0.6% versus 1.6%, OR 0.46, p = 0.001). After total hip arthroplasty 0.4% of patients developed a PJI in the vancomycin group compared to 1.8% of patients in the control group (OR 0.26, p = 0.003). After unicondylar or total knee arthroplasty, topical vancomycin led to a 0.8% rate of PJI compared to 1.8% in the control group. However, this difference failed to reach statistical significance (OR 0.55, p = 0.07). Topical vancomycin did not increase the rate of wound complications (4.5% versus 5.4%, OR 0.83, p = 0.40). There was no significant difference in overall complication rates between vancomycin and control groups (5.8% versus 7.0%, OR 0.87, p = 0.45).

The conclusions of this meta-analysis are limited by the retrospective nature of the included studies. Most studies use a consecutive series of patients without vancomycin administration followed sequentially by a series implementing topical vancomycin, or a single surgeon using vancomycin compared to a different surgeon as a control.

Additionally, results are limited by the relatively short minimum follow-up period, as many studies reported only three-month results, along with varied definitions of PJI and reporting of complications.

PJI after hip and knee arthroplasty remains a devastating and difficult to treat complication following hip and knee arthroplasty. Low level evidence suggests that topical vancomycin may be effective prophylaxis against PJI. However, given the substantial limitations of prior studies and potential for harm, higher quality studies are required before topical vancomycin can be routinely recommended. Investigators therefore propose a randomized controlled trial investigating the impact of topical vancomycin compared to standard care on PJI rates following THA and TKA.

Research Question: The overarching aim of this study is to determine whether topical vancomycin is a safe and effective intervention for the primary prevention of PJI after THA and TKA. Understanding its impact on PJI and other complication rates with high quality evidence can help make recommendations for or against its routine use and reduce risks to patients.

Study Design: The proposed research project is a pilot study which will precede a multi-centre randomized controlled trial to evaluate complication rates in THA and TKA following vancomycin administration compared to standard care. This pilot study will allow us to evaluate the study design and assess feasibility prior to implementation across Canada. Surgery will take place at one of the four major academic adult orthopedic hospitals: Peter Lougheed Center, Foothills Medical Centre, Rockyview General Hospital, and South Health Campus either Peter Lougheed Centre or Rockyview General Hospital with plans to expand to hospitals across Calgary and Canada in the future study. Investigators aim to recruit 50 patients undergoing THA and 50 patients undergoing TKA and will follow patients for one year postoperatively.

Recruitment: Initial introduction to the study will be done by the surgeons, followed by screening and recruitment, which will be completed by the research coordinator. Patients will have an opportunity to read the consent form and ask questions prior to signing the consent form. Baseline demographics including age, sex, gender, BMI, ethnicity, comorbidities, and smoking status will be recorded.

Intervention: Once enrolled, patients will be randomized preoperatively on the day of surgery Randomization will be done using R software (version 4.0.2), randomize R package. Block Randomization with randomly mixed block sizes to assign equal sample numbers to control and treatment groups (the allocator will hide the block size from the executer). This will be done via 'blockrand' Function in R. with an online randomizer (e.g. studyrandomizer.com). Patients will be blinded to their treatment arm.

Patients allocated to the control group will have all standard care infection prophylaxis interventions such as pre- and post-operative intravenous antibiotic administration, sterile surgical helmet systems, saline pulse lavage irrigation, and antimicrobial drapes. No povidone-iodine lavage will be used. Antibiotic impregnated cement may be used according to the individual surgeons' routine practices but will not differ for an individual surgeon between treatment arms.

Patients allocated to the vancomycin group will undergo all the standard care measures in addition to 1g of powdered vancomycin applied to the wound, in the intra-articular space and along wound edges after irrigation and prior to fascial closure.

Follow-up: Patients will complete follow-up at their regularly scheduled clinical follow-ups. At two weeks, six weeks, three months, six months, and one year visits patients will be assessed for the outcomes noted below.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older, who are undergoing elective primary THA or TKA for osteoarthritis
* Patients must be able and willing to complete one year of follow-up postoperatively

Exclusion Criteria:

* Patients undergoing surgery for inflammatory arthritis, post-traumatic arthritis, or avascular necrosis
* History or septic arthritis based on history or synovial aspirate
* Prior major operation on the affected joint including osteotomy, open reduction internal fixation, or major open ligamentous repair, but excluding arthroscopic procedures such as ACL reconstruction or meniscus or labral debridement/repair
* Current immunosuppressive medications
* Vancomycin allergy or history of a vancomycin-related complication such as ototoxicity or nephrotoxicity

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Periprosthetic Joint Infection in the same joint | at six weeks post-operative.
  Peri-operative Joint Infection in the operated joint
Rate of Periprosthetic Joint Infection in the same joint | at three months post-operative.
  Peri-operative Joint Infection in the operated joint
Rate of Periprosthetic Joint Infection in the same joint | at one year post-operative.
  Peri-operative Joint Infection in the operated joint

SECONDARY OUTCOMES:
Rate of reoperation | at six weeks post-operative.
  Reoperation on the same joint
Rate of reoperation | at three months post-operative.
  Reoperation on the same joint
Rate of reoperation | at one year post-operative.
  Reoperation on the same joint
Rate of superficial and non-infectious wound complications | at six weeks post-operative.
  Superficial signs of infection including erythema and warmth requiring antibiotics in the opinion of the treating physician
  * Persistent drainage lasting greater than 7 days
  * Delayed incision healing beyond 14 days
  * Seroma or hematoma requiring surgical drainage
Rate of superficial and non-infectious wound complications | at three months post-operative.
  Superficial signs of infection including erythema and warmth requiring antibiotics in the opinion of the treating physician
  * Persistent drainage lasting greater than 7 days
  * Delayed incision healing beyond 14 days
  * Seroma or hematoma requiring surgical drainage
Rate of superficial and non-infectious wound complications | at one year post-operative.
  Superficial signs of infection including erythema and warmth requiring antibiotics in the opinion of the treating physician
  * Persistent drainage lasting greater than 7 days
  * Delayed incision healing beyond 14 days
  * Seroma or hematoma requiring surgical drainage
Rate of all complications | at six weeks post-operative.
  Anaphylactic reaction
  * Ototoxicity
  * Development of laboratory confirmed antibiotic resistant organism infection or colonization
  * Acute kidney injury, defined by a serum creatine increase 1.5 times baseline
  * Blood transfusion
  * Periprosthetic fracture
  * Prosthetic dislocation
  * Radiographic osteolysis or loosening
  * Venous thromboembolism
  * Acute coronary syndrome or arrhythmia
  * Cerebrovascular accident or transient ischemic attack
  * Death
Rate of all complications | at three months post-operative.
  Anaphylactic reaction
  * Ototoxicity
  * Development of laboratory confirmed antibiotic resistant organism infection or colonization
  * Acute kidney injury, defined by a serum creatine increase 1.5 times baseline
  * Blood transfusion
  * Periprosthetic fracture
  * Prosthetic dislocation
  * Radiographic osteolysis or loosening
  * Venous thromboembolism
  * Acute coronary syndrome or arrhythmia
  * Cerebrovascular accident or transient ischemic attack
  * Death
Rate of all complications | at one year post-operative.
  Anaphylactic reaction
  * Ototoxicity
  * Development of laboratory confirmed antibiotic resistant organism infection or colonization
  * Acute kidney injury, defined by a serum creatine increase 1.5 times baseline
  * Blood transfusion
  * Periprosthetic fracture
  * Prosthetic dislocation
  * Radiographic osteolysis or loosening
  * Venous thromboembolism
  * Acute coronary syndrome or arrhythmia
  * Cerebrovascular accident or transient ischemic attack
  * Death

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Desy, MD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No